CLINICAL TRIAL: NCT06100874
Title: A Single-arm Phase II Trial of SAcituzumab Govitecan and Trastuzumab for HER2+ Metastatic Breast Cancer After Trastuzumab dEruxtEcaN (SATEEN)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adrienne G. Waks (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Adrienne G. Waks, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-531
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Her 2 Positive Breast Cancer; Breast Cancer Female; Breast Cancer Metastatic
Keywords: HER2 + Breast Cancer; HER 2 Positive Breast Cancer; Breast Cancer Female; Breast Cancer Metastatic
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Govitecan + Trastuzumab (or Biosimilar) (Experimental): Participants will complete the following:
  * Baseline visit with assessments.
  * CT or MRI scans every 9 weeks for 27 weeks and then every 12 weeks.
  * Echocardiogram or MUGA scan every 12 weeks for 24 weeks and then every 16 weeks.
  * Cycle 1 through Cycle 2:
    * Days 1 and 8 of 21 day cycle: Predetermined dose of Sacituzumab govitecan 1x daily.
    * Day 1 of 21 day cycle: Predetermined dose of Trastuzumab either intravenously or subcutaneously 1x daily.
  * Cycle 2:
    * Day 1: Optional tumor biopsy
    * Days 1 and 8 of 21 day cycle: Predetermined dose of Sacituzumab govitecan 1x daily.
    * Day 1 of 21 day cycle: Predetermined dose of Trastuzumab either intravenously or subcutaneously 1x daily.
  * Cycle 3 through End of Treatment:
    * Days 1 and 8 of 21 day cycle: Predetermined dose of Sacituzumab govitecan 1x daily.
    * Day 1 of 21 day cycle: Predetermined dose of Trastuzumab either intravenously or subcutaneously 1x daily.
  * End of treatment:
    * Follow up visits every 6 months.
  Interventions: Drug: Sacituzumab Govitecan; Drug: Trastuzumab; Drug: Trastuzumab and Hyaluronidase-oysk

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Trop-2-directed antibody-drug conjugate, 180 mg single-dose glass vial, via intravenous infusion per protocol.
  Other Names: Trodelvy
Drug: Trastuzumab — Humanized IgG1 kappa monoclonal antibody, 150mg single-dose vial, via intravenous infusion per protocol.
  Other Names: Herceptin
Drug: Trastuzumab and Hyaluronidase-oysk — Recombinant monoclonal antibody, 6 mL vial, via subcutaneous injection per protocol.
  Other Names: Herceptin Hylecta

SUMMARY:
This research study is being done to evaluate the safety and effectiveness of sacituzumab govitecan with trastuzumab (Herceptin, Herceptin Hylecta, or trastuzumab biosimilar) in metastatic HER2+ breast cancer.

The names of the study drugs used in this research study are:

* Sacituzumab govitecan (a type of antibody-drug conjugate)
* Trastuzumab (Herceptin) (a type of monoclonal antibody)
* Trastuzumab and Hyaluronidase-oysk (Herceptin Hylecta) (a type of recombinant monoclonal antibody)
* Trastuzumab biosimilar drug

DETAILED DESCRIPTION:
This is an open-label, multi-center, single-arm phase II trial to evaluate the safety and effectiveness of sacituzumab govitecan with trastuzumab (Herceptin, Herceptin Hylecta, or trastuzumab biosimilar) in metastatic HER2+ breast cancer. Participants may receive a biosimilar drug to trastuzumab, which is a nearly identical "copycat" of an original drug that is manufactured by a different company

The U.S. Food and Drug Administration (FDA) has not approved sacituzumab govitecan for Human-epidermal growth receptor 2-positive (HER2+) breast cancer, but it has been approved for triple negative breast cancer and hormone receptor positive but HER2-negative breast cancer.

The U.S. FDA has approved Trastuzumab to be administered as an IV (intravenous) or subcutaneous (injection under the skin) for HER2+ breast cancer.

The research study procedures include screening for eligibility, blood tests, Computerized Tomography (CT) scans or Magnetic Resonance Imaging (MRI) scans, biopsies, study treatment visits, echocardiograms and/or Multigated Acquisition (MUGA) scans.

It is expected that about 40 people will take part in this research study.

Gilead Sciences Inc. is supporting this research study by providing funding for the trial as well as one of the study drugs, sacituzumab govitecan.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer, with unresectable locally advanced or metastatic disease. Patients without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* At least one measurable lesion that can be accurately assessed at baseline by CT (MRI where CT is contraindicated) and is suitable for repeated assessment as per RECIST 1.149 (see Section 11).

NOTE: If the only site of measurable of disease has been previously irradiated, there must be evidence of post-radiation progression.

* Either the primary tumor or the metastasis (or both) must be HER2+ per ASCO/CAP 2018 guidelines.1 Central confirmation of HER2 status is not required.
* Any ER and PR expression are permitted but must be known.
* Participants must have received prior treatment with a taxane, trastuzumab, and T-DXd. These agents may have been administered in the curative or the advanced setting. Prior progression on these agents is not required. T-DXd does not need to be the most recent prior therapy.
* Participants must have discontinued all chemotherapy, biologic treatment or investigational agent at least 14 days prior to study treatment initiation (any prior endocrine therapy does not require washout).
* All toxicities related to prior chemotherapy must have resolved to CTCAE v5.0 grade 1 or lower, except alopecia can be any grade and neuropathy can be grade 2 or lower.
* Participants on bisphosphonates or RANK ligand inhibitors may continue receiving therapy during study treatment and also may initiate therapy with these agents on study if clinically indicated.
* Prior radiation therapy must be completed at least 7 days prior to study treatment initiation, and all toxicities related to prior radiation therapy must have resolved to CTCAE v5.0 grade 1 or lower, unless otherwise specified in 3.1.14.
* Previously treated brain metastases are permitted, with the following provisions: (1) Prior SRS should be completed ≥ 7 days before study treatment initiation; (2) Prior WBRT should be completed ≥ 7 days before study treatment initiation. (3) Any corticosteroid use for brain metastases must have been discontinued for ≥ 7 days prior to study treatment initiation.
* Pre- and postmenopausal women or male patients ≥ 18 years old.
* ECOG performance status of 0 - 2 (Karnofsky > 50%).
* Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
* Participants must have normal organ and bone marrow function as defined below:

  * Absolute neutrophil count ≥1,000/mcL
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥ 9.0 g/dl
  * INR/PT/aPTT ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is in therapeutic range of anticoagulant
  * Total bilirubin ≤1.5 × institutional upper limit of normal (ULN) (or ≤2.0 x ULN in patients with documented Gilbert's Syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN or

    ≤5 × institutional ULN for participants with documented liver metastases
  * Serum creatinine ≤1.5 × institutional ULN OR creatinine clearance ≥ 30 mL/min/ 1.73m2 for participants with creatinine levels above institutional ULN.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 2 weeks prior to study treatment initiation. Childbearing potential is defined as participants who have not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and have not undergone surgical sterilization (removal of ovaries and/or uterus).
* WOCBP must agree to use an adequate method of contraception. Contraception is required starting with the first dose of study medication through 7 months after the last dose of study medication. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormone-releasing intrauterine devices, and copper intrauterine devices. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception (Appendix C).
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment 7 months after the last dose of study treatment.
* Participants must be willing to undergo a research biopsy at baseline. If disease is not safely accessible according to the treating investigator, permission to waive the mandatory baseline biopsy must be received from the sponsor-investigator. Patients must be willing to provide archival tissue for research purposes.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior therapy with any Trop-2 directed ADC, including sacituzumab govitecan.
* Prior hypersensitivity to trastuzumab, sacituzumab govitecan, or the excipients of trastuzumab or sacituzumab govitecan.
* Known history of UDP-glucuronosyltransferase 1A1 (UGT1A1) *28 allele homozygosity, which is associated with increased risk for neutropenia and diarrhea related to irinotecan.50 UGT1A1 genotyping is not required for eligibility.

Note: Concurrent administration of strong UGT1A1 inhibitors or inducers is not allowed during the study (See Section 5.5).

* Known brain metastases that are untreated, symptomatic, or require corticosteroid therapy to control symptoms.
* Known leptomeningeal disease.
* Major surgery within 2 weeks prior to study treatment initiation. Patients must have recovered from any effects of any recent major surgery.
* Individuals with a history of a second malignancy are ineligible except for the following circumstances:

  * Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the investigator to be at low risk for recurrence of that malignancy.
  * Individuals with the following cancers that have been diagnosed and treated within the past 3 years are eligible: cervical/prostate carcinoma in situ, superficial bladder cancer, non-melanoma cancer of the skin.
  * Patients with other cancers diagnosed within the past 3 years and felt to be at low
  * risk of recurrence should be discussed with the study principal investigator to determine eligibility.
* Uncontrolled, significant intercurrent or recent illness including, but not limited to, ongoing or active infection, uncontrolled non-malignant systemic disease, uncontrolled seizures, or psychiatric illness/social situation that would limit compliance with study requirements in the opinion of the treating investigator.
* Participants who are pregnant or breast-feeding are not eligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 3 years
  The overall response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECISTv1.1 criteria.

SECONDARY OUTCOMES:
Median Progression-Free Survival (PFS) | 3 years
  Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last disease assessment.
Median Overall Survival (OS) | 10 years
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Clinical Benefit Rate (CBR) | 3 years
  CBR defined as proportion of participants with Partial Response (PR) + Complete Response (CR) + Stable Disease (SD) ≥6 months per RECIST 1.1
Median Duration of Overall Response (DOR) | 3 years
  Duration of Overall Response (DOR), estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) per RECISTv1.1, until the first date that recurrent or progressive disease is objectively documented. Patients without progressive disease are censored at the date of last disease assessment.
Grade 3-5 Treatment-related Toxicity Rate | 3 years
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Waks, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Miami Cancer Institute at Baptist Health, Miami, Florida
  - Dana Farber Cancer Institite, Boston, Massachusetts
  - DFCI @ South Shore Hospital, South Weymouth, Massachusetts
  - SCRI Oncology Partners, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu